CLINICAL TRIAL: NCT03750006
Title: Enhancing Functional Capacity in Older Adults With Short Session High Intensity Interval Training
Acronym: HIIT-VA
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: COVID pandemic halted ability to enroll participants. Grant funded then ended.
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Collaborators: The VA Western New York Healthcare System (U.S. Federal Agency); University at Buffalo (Other); Roswell Park Cancer Institute (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: E2902-P; RX002902 (Other Grant/Funding Number: Veteran Affairs)
Record Dates: First submitted 2018-11-09; First posted 2018-11-21 (Actual); Results first posted 2024-08-30 (Actual); Last update posted 2024-08-30 (Actual); Status verified 2024-08

CONDITIONS: Frailty
Keywords: frailty; sarcopenia; exercise; high intensity; older adults; microRNA
MeSH Terms: conditions — Frailty; Sarcopenia; Motor Activity

STUDY DESIGN:
Intervention Model Description: The goals of this proposal are to: 1) investigate the feasibility of recruiting and administering short session HIIT to frail, pre-frail, and non-frail older Veterans and 2) to characterize the physical performance benefits and serum microRNA (miRNA) profiles in those participants.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- HIIT intervention (Experimental): Individually tailored short session high intensity interval training session 3 times per week for 12 weeks on a recumbent exercise cycle.
  Interventions: Behavioral: Short session HIIT

INTERVENTIONS:
Behavioral: Short session HIIT — Individually tailored short session high intensity interval training session 3 times per week for 12 weeks on a recumbent exercise cycle.

SUMMARY:
Frailty is a clinical condition of poor physiological reserve that increases risks for adverse health outcomes including falls, hospitalization and mortality. Exercise is beneficial for the prevention and even reversal of frailty, yet participation among older individuals is limited. Short session high intensity interval training (HIIT) is emerging as a promising exercise strategy that achieves performance gains with lower time commitment. The goal of this pilot proposal is to establish the feasibility of HIIT exercise training protocols in 65-85 year old individuals, as well as to demonstrate the ability to detect functional and physiologic benefits. The investigators anticipate the preliminary research findings will lay the foundation for future human clinical studies that will permit us to significantly improve the health of Veterans.

DETAILED DESCRIPTION:
Enhancing functional capacity in older adults with short session high intensity interval training

Frailty is a condition of poor physiological reserve that increases susceptibility to falls, hospitalization, disability and mortality. The incidence of frailty rapidly increases after the age 65, growing from 10% to as many as 50% of those 85 years or older; therefore over 9 million Veterans are either frail or at risk for frailty. Exercise has proven benefits for frailty, yet older adults rarely attain the recommended 150 minutes a week of moderate intensity exercise. High intensity interval training (HIIT) is emerging as an alternative as it delivers similar or better gains than moderate intensity exercise in less time. Recently, the investigators published that a 3-day-a-week, 10-minute HIIT regimen in aged mice not only reduces frailty, but leads to both strength and endurance benefits. In addition, the preliminary data demonstrate significant changes in microRNA (miRNA) profiles. Despite the potential of short session HIIT to improve functional capacity and lead to better adherence, the modality has not been tested in individuals 65-85 years of age, and in particular, frail individuals. The goals of this proposal are to: 1) investigate the feasibility of recruiting and administering short session HIIT to frail, pre-frail, and non-frail older Veterans and 2) to characterize the physical performance benefits and serum microRNA (miRNA) profiles in those participants.

To accomplish these goals the investigators will administer a short session HIIT regimen totaling only 10-minutes, 3-days-a-week for 3 months, using recumbent exercise cycles, to 65-85 year old participants. The investigators will also utilize next generation RNA sequence technology to assess HIIT impacts upon microRNA profiles in serum samples. The investigators anticipate this project will demonstrate the feasibility of administering short session HIIT to older individuals, including vulnerable frail and pre-frail populations as well as demonstrate the ability to collect and analyze serum miRNA profiles. The advantages to this program are the ability to maintain or build muscle mass and improve aerobic conditioning, especially in older patients where frailty and sarcopenia are so prevalent. This pilot project will therefore lay the foundation for future clinical trials that further explore the utility of HIIT to prevent or delay the onset of frailty in larger cohorts, and ultimately lead to the enhancement of functional capacity and quality of life in aging Veteran populations.

ELIGIBILITY:
Inclusion Criteria:

* Male or female
* Any race
* Frail, pre-frail, and non-frail
* Medical clearance for exercise

Exclusion Criteria:

* Severe co-morbidity (e.g. - CHF (class III), COPD (GOLD stage IV), CKD (stage 3))
* VAMC SLUMS score 20
* Physical impairment that prevents use of a recumbent exercise bike

Ages: 60 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2018-12-03 (Actual); Primary Completion 2021-12-31 (Actual); Study Completion 2022-12-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bruce R. Troen, MD, Principal Investigator — VA Western New York Healthcare System, Buffalo, NY
Locations (1):
- VA Western New York Healthcare System, Buffalo, NY, Buffalo, New York, United States

IPD SHARING:
Plan to Share IPD: Yes
Thus, the investigators will make the data and associated documentation available to users only under a data-sharing agreement that provides for: (a) a commitment to using the data only for research purposes and not to identify any individual participant; (b) a commitment to securing the data using appropriate computer technology; (c) restrictions on redistribution of the data to third parties, and proper acknowledgement of the data resource, and (d) a commitment to destroying or returning the data after analyses are completed. De identified data will be maintained on a VA server and will only be shared via encrypted devices. Co-Investigators will have access to the data collected as part of their aims. Investigators working on the grant will have access to the data through the PI. The data will be monitored routinely to maintain safety and productivity, as well as to assist with research dissemination annually.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: Six months after publication.
Access Criteria: Final data sets will be made available upon specific request and under an authorized Data Use Agreement. This, in addition to the publications being made available via PubMed Central, will enable validation of results by recipients.

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment from 12/3/2018 - 12/31/2019. Recruitment occurred at the VA Western New York including through posted advertisements and word of mouth.
Pre-assignment Details: 11 individuals were excluded due to the COVID pandemic.
Period: Overall Study
Arm/Group | HIIT Intervention
Started (Recruitment initiated) | 42
Completed | 23
Not Completed | 19
Not completed — Withdrawal by Subject | 8
Not completed — COVID PANDEMIC | 11

BASELINE CHARACTERISTICS:
Arm/Group | HIIT Intervention
Number analyzed (Participants) | 23
Age, Continuous [Mean (Standard Deviation); unit: years] | 71.9 (6.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1
  Male | 22
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 23
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 4
  White | 19
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 23
BMI [Mean (Standard Deviation); unit: kg/m^2] | 30.6 (0.6076)
Smoking status [Count of Participants; unit: Participants]
  Non-smoker | 5
  Former Smoker | 16
  Current Smoker | 2

OUTCOME MEASURES:

1. Primary Outcome: 6-minute Walk at Baseline and Endpoint
Description: 6-minute walk, total distance over 6 minutes in a 50 foot long hallway, participants asked to walk at a "brisk" pace.
Time Frame: baseline and at participant completion, an average of 3 months
Measure: Mean (Standard Deviation); unit: meters
Arm/Group | HIIT Intervention
Number analyzed (Participants) | 23
meters
  Baseline | 418.2 (72.2)
  Endpoint | 436.8 (55.6)
Statistical Analysis 1: Comparison: HIIT Intervention; Test type: Superiority; p = 0.0238, t-test, 2 sided — Not adjusted for multiple comparisons, P < 0.05 is considered significant; paired T-test

2. Primary Outcome: Physical Activity Enjoyment at Baseline and Endpoint
Description: Physical Activity Enjoyment Scale (PACES) that provides a valid instrument for assessing enjoyment in physical activity. There are 18 questions, each of which can receive a score from 1 to 7, where 7 is represents greater enjoyment. Scores presented as the mean across all questions giving an overall range of 1-7.
Time Frame: baseline and at participant completion, an average of 3 months
Population: One participant was not able to complete the assessment due to scheduling conflict.
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | HIIT Intervention
Number analyzed (Participants) | 22
Scores on a scale
  Baseline | 6.1 (0.8)
  Endpoint | 6.2 (0.8)
Statistical Analysis 1: Comparison: HIIT Intervention; Test type: Superiority; p = 0.3029, t-test, 2 sided; Paired, P < 0.05 is considered significant

3. Primary Outcome: VO2max at Baseline and Endpoint
Description: Performed as part of a symptom limited maximal endurance test on a cycle ergometer
Time Frame: baseline and at participant completion, an average of 3 months
Population: 8 participants were not able to complete the VO2max end point assessment due to COVID pandemic study cessation.
  One participant was not able to complete the assessment due to scheduling conflict.
Measure: Mean (Standard Deviation); unit: mL/min/kg
Arm/Group | HIIT Intervention
Number analyzed (Participants) | 14
mL/min/kg
  Baseline | 18.67 (5.12)
  Endpoint | 19.93 (5.59)
Statistical Analysis 1: Comparison: HIIT Intervention; Test type: Superiority; p = 0.1713, t-test, 2 sided; Paired, P < 0.05 is considered significant

4. Secondary Outcome: Short Physical Performance Battery at Baseline and Endpoint
Description: Short Physical Performance Battery (SPPB) is an objective assessment tool for evaluating lower extremity functioning in older persons, including balance, side-by-side/semi-tandem/tandem stands, and gait speed. There are 3 subscales, each of which can receive from 0 to 4 points. Therefore the total range of the test spans summed scores from 0 to 12, where 12 is the best outcome.
Time Frame: baseline and at participant completion, an average of 3 months
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | HIIT Intervention
Number analyzed (Participants) | 23
score on a scale
  Baseline | 10.11 (2.0)
  Endpoint | 10.46 (2.1)
Statistical Analysis 1: Comparison: HIIT Intervention; Test type: Superiority; p = 0.1261, t-test, 2 sided; paired, P < 0.05 is considered significant

5. Secondary Outcome: Frailty at Baseline and Endpoint
Description: Fried frailty phenotype assessment includes: gait speed, grip strength, endurance, activity level, weight loss.
  These assessments report summed scores of 0 to 5, where 0 is the best outcome. If gait speed or grip strength (m/sec or kg) falls within the lowest quintile (20%) for the age and gender adjusted range, then it is given a score of "1". If both questions on the endurance or activity measures are positive then then it is given a score of "1". If weight loss is greater than 5% over the past year, then it is given a score of "1".
Time Frame: baseline and at participant completion, an average of 3 months
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | HIIT Intervention
Number analyzed (Participants) | 23
score on a scale
  Baseline | 0.87 (0.8)
  Endpoint | 0.61 (0.8)
Statistical Analysis 1: Comparison: HIIT Intervention; Test type: Superiority; p = 0.1367, t-test, 2 sided; paired, P < 0.05 is considered significant

6. Secondary Outcome: Quality of Life Survey at Baseline and Endpoint
Description: Quality of Life Enjoyment and Satisfaction Questionnaire - Short Form (Q-LES-Q-SF). There are 14 subscales with scores of 1 to 5, where 5 is the better outcome. Therefore the total range of the test spans scores from 14 to 70, where 70 is the best outcome. The final score as a percentage with range being 0-100% and top being 100%. This percentage is calculated as: 100 * ((participant's score - 14) / 56).
Time Frame: baseline and at participant completion, an average of 3 months
Measure: Mean (Standard Deviation); unit: % of Max Score
Arm/Group | HIIT Intervention
Number analyzed (Participants) | 23
% of Max Score
  Baseline | 80.0 (11.4)
  Endpoint | 85.6 (9.6)
Statistical Analysis 1: Comparison: HIIT Intervention; Test type: Superiority; p = 0.0111, t-test, 2 sided; paired, P < 0.05 is considered significant

7. Secondary Outcome: Cognitive Survey at Baseline and Endpoint
Description: VA-SLUMS: VA Saint Louis University Mental Status screen. Survey includes 11 questions allowing a range of scores from 1-30 points, where higher scores represent greater mental outcomes.
Time Frame: baseline and at participant completion, an average of 3 months
Population: One participant was not able to complete the assessment due to scheduling conflict.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | HIIT Intervention
Number analyzed (Participants) | 22
score on a scale
  Baseline | 26.6 (2.5)
  Endpoint | 27.3 (2.3)
Statistical Analysis 1: Comparison: HIIT Intervention; Test type: Superiority; p = 0.0219, t-test, 2 sided; Paired, P < 0.05 is considered significant

8. Secondary Outcome: Activities of Daily Living & Instrumental Activities of Daily Living Survey at Baseline and Endpoint
Description: The Activities of Daily living and instrumental activities of daily living are a survey comprised of 14 questions including ability to: dress, eat, ambulate, toilet, hygiene, shop, housework, accounting, food preparation, and use transportation/telephone. Each question gives up to 1 point with a total range of 0-14. Higher scores indicate less independence and greater reliance on support.
Time Frame: baseline and at participant completion, an average of 3 months
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | HIIT Intervention
Number analyzed (Participants) | 23
Score on a scale
  Baseline | 0.04 (0.21)
  Endpoint | 0.0 (0.0)
Statistical Analysis 1: Comparison: HIIT Intervention; Test type: Superiority; p = 0.3660, t-test, 2 sided; Paired, P < 0.05 considered significant

9. Secondary Outcome: microRNA Profiling at Baseline and Endpoint
Description: Next Generation Sequencing of microRNA species from serum.
Time Frame: baseline and at participant completion, an average of 3 months
Population: RNA was isolated from participant serum samples and sequenced. However, none of the sequenced RNA were microRNA sequences, therefore analysis could not be performed. Consequently, there was no microRNA data that could be presented in a table.
Arm/Group | HIIT Intervention
Number analyzed (Participants) | 0

10. Secondary Outcome: Serum 25-hydroxy-vitamin D at Baseline
Description: serum 25-hydroxy-vitamin D was measured from serum isolated from blood collected at baseline and measured using ELISA
Time Frame: baseline
Population: No Statistical Analysis was performed as this was only a baseline measurement.
Measure: Mean (Standard Deviation); unit: ng/ml
Arm/Group | HIIT Intervention
Number analyzed (Participants) | 23
ng/ml | 26.9 (15.2)

11. Secondary Outcome: C-reactive Protein Level at Baseline and Endpoint
Description: C-reactive protein was measured from isolated serum samples at baseline and endpoint using ELISA
Time Frame: baseline and at participant completion, an average of 3 months
Measure: Mean (Standard Deviation); unit: ug/uL
Arm/Group | HIIT Intervention
Number analyzed (Participants) | 23
ug/uL
  Baseline | 3.0 (3.5)
  Endpoint | 3.7 (3.7)
Statistical Analysis 1: Comparison: HIIT Intervention; Test type: Superiority; p = 0.1563, t-test, 2 sided; Paired, P < 0.05 is considered significant

12. Secondary Outcome: Quadriceps Strength at Baseline and Endpoint
Description: Maximal quadriceps strength. This will be measured with the MicroFET2 dynamometer with a readout in kilograms (kg) of force.
Time Frame: baseline and at participant completion, an average of 3 months
Population: One participant was not able to complete the assessment due to scheduling conflict.
Measure: Mean (Standard Deviation); unit: kg
Arm/Group | HIIT Intervention
Number analyzed (Participants) | 22
kg
  Right Leg - Baseline | 27.7 (6.8)
  Right leg - Endpoint | 31.1 (7.1)
  Left leg - Baseline | 28.0 (7.9)
  Left Leg - Endpoint | 29.9 (6.9)
Statistical Analysis 1: Comparison: HIIT Intervention; Test type: Superiority; p = 0.0110, t-test, 2 sided; Paired, P < 0.05 is considered significant

13. Secondary Outcome: FRAIL Scale Survey at Baseline and Endpoint
Description: FRAIL scale: fatigability, resistance, ambulation, illnesses, loss of weight. If the answers to any of the questions is yes, then given score is "1" with a total survey range of 0 to 5. Higher scores represent greater frailty.
Time Frame: baseline and at participant completion, an average of 3 months
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | HIIT Intervention
Number analyzed (Participants) | 23
Score on a scale
  Baseline | 0.2 (0.4)
  Endpoint | 0.1 (0.3)
Statistical Analysis 1: Comparison: HIIT Intervention; Test type: Other; p = 0.3282, t-test, 2 sided; Paired, P < 0.05 is considered significant

14. Secondary Outcome: Serum Interleukin-6 Level at Baseline and Endpoint
Description: Interleukin-6 collected from serum extracted from blood samples taken at baseline and endpoint and measured using ELISA
Time Frame: baseline and at participant completion, an average of 3 months
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | HIIT Intervention
Number analyzed (Participants) | 23
pg/mL
  Baseline | 3.8 (1.9)
  Endpoint | 4.2 (2.4)
Statistical Analysis 1: Comparison: HIIT Intervention; Test type: Superiority; p = 0.5244, t-test, 2 sided; Paired, P < 0.05 is considered significant

15. Secondary Outcome: Serum Interleukin-10 Level at Baseline and Endpoint
Description: Interleukin-10 collected from serum extracted from blood samples taken at baseline and endpoint and measured using ELISA
Time Frame: baseline and at participant completion, an average of 3 months
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | HIIT Intervention
Number analyzed (Participants) | 23
pg/mL
  Baseline | 3.0 (0.9)
  Endpoint | 3.1 (1.2)
Statistical Analysis 1: Comparison: HIIT Intervention; Test type: Superiority; p = 0.5718, t-test, 2 sided; Paired, P < 0.05 is considered significant

16. Secondary Outcome: Number of Participants With Muscle Tissue Oxygenation Raw Data Collected
Description: Seeking to collect raw data using functional near infra-red spectroscopy to analyze quadriceps during VO2max test. This work is the first steps in the development of techniques that analyze muscle blood flow and tissue oxygenation during exercise.
Time Frame: baseline and at participant completion, an average of 3 months
Population: The goal of this project was to determine if raw functional near infrared spectroscopy data could be collected in participants. Data collection was verified. This work lays the foundation for future efforts in new experiments to determine methods to analyze the raw data to generate understandable data for interpretation - and lead to better understanding of the impacts of exercise on blood flow in muscle tissue.
Measure: Count of Participants; unit: Participants
Arm/Group | HIIT Intervention
Number analyzed (Participants) | 23
Participants | 10

ADVERSE EVENTS:
Time Frame: Adverse event data were collected weekly over a 14 week period for each participant, commencing from baseline assessments week 0, through the HIIT intervention (weeks 1 - 12 or up to 14), and ending with collection at end-point assessments.
Arm/Group | HIIT Intervention
All-Cause Mortality (participants affected / at risk) | 0/23
Serious Adverse Events (participants affected / at risk) | 0/23
Other Adverse Events (participants affected / at risk) | 0/23

LIMITATIONS AND CAVEATS:
Goal of trial was to evaluate recruitment, administration, and safety profile of short session HIIT, and not necessarily the efficacy of the HIIT protocol for functional capacity.

Trial does not have a non-exercise control group Trial features limited number of participants (23), which includes only 1 female Trial was stopped short due to COVID-19 pandemic, 8 of the 23 participants did not complete the total 12 weeks of training although all participants had at least 6 weeks of training.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2022-01-25): https://cdn.clinicaltrials.gov/large-docs/06/NCT03750006/Prot_SAP_000.pdf
  • Informed Consent Form (2021-11-17): https://cdn.clinicaltrials.gov/large-docs/06/NCT03750006/ICF_001.pdf